CLINICAL TRIAL: NCT02033304
Title: Analysis of Factors Predicting Postoperative Pain and Wound Hyperalgesia After Cesarean Section
Brief Title: Factors Predicting Postoperative Cesarean Section Pain
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 7124
Record Dates: First submitted 2014-01-09; First posted 2014-01-10 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2013-01

CONDITIONS: Postoperative Pain
Keywords: Cesarean section; Pain; Wound hyperalgesia
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In spite of identical analgesic protocols, parturients suffer different levels of pain postoperative lay. In this study we hope to identify factors which influence the perception of pain including preoperative anxiety, sleep quality and local anesthesia injection pain.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing spinal anesthesia

Exclusion Criteria:

* women unable to cooperate
* Women undergoing general anesthesia

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women after cesarean section
Sampling Method: Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | Postoperative day1

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Beilinson hospital, Petach Tikvah
  - Rabin medical center, Petach Tikvah